CLINICAL TRIAL: NCT05001906
Title: Research on the Influence of Prenatal Exercise on Circulatory Function and Structure of Pregnant Women
Brief Title: Pregnant Women With Physical Activity
Acronym: GineVeiw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Banja Luka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EO2619
Record Dates: First submitted 2021-07-19; First posted 2021-08-12 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-05

CONDITIONS: Pregnancy
Keywords: Pregnancy; Physical exercise; Cardiovascular system; Gestational weight gain
MeSH Terms: conditions — Motor Activity; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group (CG) will consist of pregnant women with standard prenatal care, who attending theoretical classes on childbirth (CG, n = 35). The control group will not exercise. The sedentary participants will continue their regular daily activities and life habits.
- Exercise group (Experimental): The exercise group (EG) will consist of pregnant women who will attend theoretical classes and prenatal exercises in the program of psychophysical preparation for childbirth (EG, n = 35). The experimental group will exercise for 45 minutes, three times a week.
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — The exercise program comprises static and dynamic breathing exercises, muscle stretching exercises and muscle strength exercises, exercises to strengthen the abdominal wall muscles, exercises to strengthen the thigh muscles - quadriceps femoris (lat. musculus quadriceps femoris), to strengthen gluteal muscles, exercises to increase pelvic mobility, exercise to improve circulation, as well as pelvic floor muscle training with relaxation techniques.
  Arms: Exercise group

SUMMARY:
Physical activity, defined as any movement of the body produced by the contraction of skeletal muscles in all phases of life, maintains and improves cardiorespiratory capacity, reduces the risk of obesity and associated comorbidities. The study will analyze the effect of prenatal exercise on circulatory functional and structural parameters and gestational weight gain in pregnant women who exercised regularly, compared to pregnant women who did not exercise regularly.

DETAILED DESCRIPTION:
Physical activity, defined as any movement of the body produced by the contraction of skeletal muscles in all phases of life, maintains and improves cardiorespiratory capacity, reduces the risk of obesity and associated comorbidities. The incidence of a sedentary lifestyle during pregnancy ranges from 64.5 to 91.5% and tends to increase in the third trimester. This has a negative impact on the quality of life and contributes to the obesity epidemic in pregnant women. Physical inactivity and excessive weight gain during pregnancy increase the risk of gestational diabetes and pregnancy-induced hypertension. In pregnancy, the circulatory system adapts to adequately supply the needs of the mother and fetus. Physical activity is considered a preventive measure for the diseases of the cardiovascular system in pregnancy.

The study will analyze the effect of prenatal exercise on circulatory functional and structural parameters and gestational weight gain in pregnant women who exercised regularly, compared to pregnant women who did not exercise regularly.

In the first phase of the study, an experimental and control group will be formed. The prenatal exercise program will be conducted with the experimental group for 8 weeks. The control group will not exercise, will have standard prenatal care, and attend classes of theoretical classes on childbirth. Respondents in both groups will fill out a questionnaire from which the data will be obtained: age, height, bodyweight before pregnancy. Data on the week of pregnancy will be obtained from the medical documentation.

The prenatal exercise program was made according to the recommendations of the American College of Obstetricians and Gynecologists (ACOG recommendations) and the guidelines of the Croatian Association of Physiotherapists for Women's Health.

The exercise program is presented with: muscle stretching exercises and muscle strength exercises, exercises to strengthen the abdominal wall muscles, exercises to strengthen the thigh muscles - quadriceps femoris (lat. musculus quadriceps femoris), to strengthen gluteal muscles, exercises to increase pelvic mobility, exercise to improve circulation, as well as pelvic floor muscle training with breathing and relaxation techniques.

Bodyweight will be measured at the beginning of the test, at the end of the exercise program, and at the end of the pregnancy.

Blood pressure data will be obtained by measuring blood pressure with a mercury manometer with a mercury column, in both groups: at the beginning of the study and the end of the study.

The shape of capillary loops and the number of capillary loops of the nail skin fold will be analyzed with nailfold capillaroscopy in both groups of subjects: at the beginning of the study and after 8 weeks.

In the second phase of the work, the collected data will be processed by methods of descriptive and parametric statistics.

The obtained results will be presented at the third phase of the work.

ELIGIBILITY:
Inclusion Criteria:

* age of pregnant women from 20 to 40 years
* a normal pregnancy confirmed by a gynecologist
* duration of pregnancy from the 20th to the 32nd gestational week
* body mass index (BMI) before pregnancy <25 kg/m2
* single pregnancy.

Exclusion Criteria:

* bleeding in the second or third trimester
* premature birth in the current pregnancy,
* rupture of the amniotic sac,
* preeclampsia or pregnancy-induced hypertension,
* intrauterine growth restriction (IUGR) in the current pregnancy,
* anemia
* not being regular in the physical exercise program
* at the pregnant woman's own request.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure at time point 1 | 20-32 weeks of gestation
  The blood pressure of pregnant women would be measured using a standard mercury manometer and compared in between study groups. In the experimental group, blood pressure would be measured at the beginning of prenatal exercises, between 20 and 32 weeks of gestation. In the control group, blood pressure would be measured at the beginning of theoretical classes, between 20 and 32 weeks of gestation.
Systolic and diastolic blood pressure at time point 2 | 28-40 weeks of gestation
  Using a standard mercury manometer blood pressure would be measured in the experimental group after eight weeks of prenatal exercises (between 28 and 40 weeks of gestation) and in the control group after eight weeks of theoretical classes (between 28 and 40 weeks of gestation).

SECONDARY OUTCOMES:
Gestational weigh gain | 38 weeks pregnancy
  Weight gain during pregnancy measured in kilograms would be determined.
Shape of nailfold capillary loops | 20-32 weeks and 28-40 weeks gestation
  The shape of capillary loops of the nail skin fold would be assessed with nailfold capillaroscopy at the beginning of prenatal exercises, between 20 and 32 weeks of gestation, and at the end of prenatal exercises, between 28 and 40 weeks of gestation.
Nailfold capillary density | 20-32 weeks and 28-40 weeks gestation
  The density of capillary loops of the nail skin fold would be assessed as the number of capillary loops per 1 mm of the distal row of capillary in nailfold (capillary/mm). The measurements will be realized at the beginning of prenatal exercises, between 20 and 32 weeks of gestation, and at the end of prenatal exercises, between 28 and 40 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Ljubojevic, MD PhD, Study Chair — Faculty of Medicine, University of Banja Luka; Vlatka Bojanic, MSN, Principal Investigator — Faculty of Medicine, University of Banja Luka
Locations (1):
- University of Banja Luka, Faculty of Medicine, Banja Luka, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Data that will be shared are individual participant data that underlie the results reported in the article (text, tables, figures)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available 3 months following publication and ending 36 months following article publication.
Access Criteria: Proposals should be directed to vesna.ljubojevic@med.unibl.org.The proposal may be submitted up to 36 months following article publication.